CLINICAL TRIAL: NCT06558578
Title: Association of Helicobacter Pylori Infection and Migraine in Children and Adolescent
Brief Title: Association of Helicobacter Pylori Infection and Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ragab Ali, Principal investigator, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: soh-Med-27-07-14MS
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Migraine in Children
MeSH Terms: interventions — Defecation; Endoscopy, Digestive System

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator): Children with migraine (cases) Inclusion criteria Age: children between 6 and 16 years old. Both sexes. children who suffering from migraine.
  Exclusion criteria:
  Age: children below 6 years old& children above 16 years old. Children suffering from epilepsy, Mental retardation, autism, attention deficient hyperactivity disorder.
  Interventions: Diagnostic Test: Helicobacter pylori antigen in stool
- Control (Other): Healthy children (control) healthy children not suffering from migraine or any neurological diseases.
  Interventions: Diagnostic Test: Helicobacter pylori antigen in stool

INTERVENTIONS:
Diagnostic Test: Helicobacter pylori antigen in stool — H pylori antigen in stool: for all patients suffering from migraine and control group.
  Upper GIT endoscopy: for children with positive H Pylori antigen in stool.
  Other Names: Upper gastrointestinal tract endoscopy

SUMMARY:
The study aims to assess the relation between migraine and H pylori infection in children and adolescent.

DETAILED DESCRIPTION:
Migraine is one of the most common types of headaches worldwide, affecting 12-15% of the world population, more common in women and also the main headache for which patients refer to specialist nerve clinics.

Migraine is a complex neurovascular condition involving vasodilatation of intracranial and extracerebral blood vessels. This results in activation of trigeminal sensory nervous pain pathway leading to headache. Serotonin and reserpine (serotonin evacuator) play a notable role in the development of migraine headache by increasing cerebral blood flow.

Migraine is characterized by episodic attack that may be moderate to severe in intensity, focal in nature, have a throbbing quality. Compared to adults, pediatric migraine is shorter in duration and often has bilateral, bifrontal in the point of location.

Migraine is divided into two main types of migraine are: migraine with aura in which patients experience transient visual or sensory symptoms (including flickering lights, spots, or pins that develop 5-20 minutes before attacks), occurring in approximately 25% of patients with migraine, and migraine without aura, occurring in the remaining 75% of patients .

Helicobacter pylori infection is a significant risk factor for migraine with no observational difference between two types (migraine with and without aura). Eradication treatment was helpful on the clinical improvement of pain.

H. pylori is a gram-negative, microaerophilic, spiral bacterium with increased motility by multiple unipolar flagella. It generates urease and colonizes the mucus layer adjacent to the gastric mucosa, usually being responsible for gastrointestinal impairments such as chronic active gastroenteritis, infection, gastric and duodenal ulcer, and, more rarely, stomach cancer, also may be the result of various extra-digestive conditions such as neurological, cardiovascular, metabolic, hematologic, ocular, or dermatological ones.

A research explained that gastrointestinal neuroendocrine cells such as enterochromaffin cells (EC cells) can synthesize and secrete serotonin (5-hydroxytryptamine; 5-HT) and some factors that motivate the cell to secrete 5-HT can cause central nervous system (CNS) perturbation via the brain-gut axis. Inflammation motivates the cell to secrete 5-HT e.g., when H. pylori infect a cell. Eradication of H. pylori infection has helpful outcomes to improve clinical attacks by the effect of eradication therapy on the inflammation induced high levels of 5-HT .

Other theory suggests that during the infection, superoxide radicals and NO are produced and prolonged oxidative injury caused by the persistent infection might be involved in regional cerebral flow changes during migraine .

ELIGIBILITY:
-Inclusion criteria: children between 6 and 16 years old. Both sexes. children who suffering from migraine.

-Exclusion Criteria: children below 6 years old& children above 16 years old. Children suffering from epilepsy, Mental retardation, autism, attention deficient hyperactivity disorder.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
migraine in children and adolescent | Over 1 year
  assessment the association between migraine and H pylori infection in children and adolescent.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ragab, Principal Investigator — Mohamed Ragab
Locations (1):
- Faculty of medicine sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No